CLINICAL TRIAL: NCT00079014
Title: A Phase I Study of Triapine® in Combination With Doxorubicin in Refractory Tumors
Brief Title: 3-AP and Doxorubicin In Treating Patients With Metastatic or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00011; CO 03904; WCCC-CO-03904; NCI-6266; P30CA014520 (NIH); U01CA062491 (NIH)
Record Dates: First submitted 2004-03-08; First posted 2004-03-09 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — 3-aminopyridine-2-carboxaldehyde thiosemicarbazone; Doxorubicin

ARMS (1):
- Treatment (triapine, doxorubicin hydrochloride) (Experimental): Patients receive doxorubicin IV over 15 minutes on day 1 and 3-AP (Triapine®) IV over 2 hours on days 1-4. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of 3-AP (Triapine®) until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, an additional 6 patients are treated at that dose level.
  Interventions: Drug: triapine; Drug: doxorubicin hydrochloride; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: triapine — Given IV
  Other Names: 3-AP; OCX-191
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects and best dose of 3-AP and doxorubicin in treating patients with metastatic or refractory solid tumors. Drugs used in chemotherapy, such as doxorubicin, work in different ways to stop tumor cells from dividing so they stop growing or die. 3-AP may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth and may help doxorubicin kill more cancer cells by making them more sensitive to the drug.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To find the maximal tolerated dose for the combination of doxorubicin and Triapine® in patients with refractory solid tumors.

SECONDARY OBJECTIVES:

I. To find the severity and frequency of toxicity associated with this combination and to observe for and record any antitumor activity.

TERTIARY OBJECTIVES:

I. To evaluate the effect of Triapine®/doxorubicin on the ribonucleotide reductase tyrosyl radical in vivo by EPR spectroscopy in buccal mucosal cells, peripheral blood lymphocytes and in tumor biopsies. Formation of low molecular weight iron-Triapine® chelates will also be assessed by EPR.

II. To evaluate the effect of Triapine®/doxorubicin on cell cycle in vivo by measuring S-phase arrest in buccal mucosal cells.

III. To evaluate the effect of Triapine®/doxorubicin on MDR gene expression and polymorphisms in blood.

IV. To evaluate the effect of Triapine®/doxorubicin on ribonucleotide reductase R2 mRNA and immunohistochemistry.

V. To evaluate the pharmacokinetic profile of the combination. VI. To measure the formulation of circulating isoprostanes as an indicator of oxidative stress with this combination.

OUTLINE: This is a dose-escalation study of 3-AP (Triapine^®).

Patients receive doxorubicin IV over 15 minutes on day 1 and 3-AP (Triapine®) IV over 2 hours on days 1-4. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of 3-AP (Triapine®) until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, an additional 6 patients are treated at that dose level.

Patients are followed until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative chemotherapy measures do not exist or are no longer effective
* Patients must not have previously received anthracyclines
* Patients must not have received radiation to > 25% of bone marrow
* ECOG performance status =< 2
* Life expectancy of greater than 12 weeks
* Leukocytes >= 3,000/μl
* Absolute neutrophil count >= 1,500/μl
* Platelets >= 100,000/μl
* Total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT) =< 2.5 X institutional upper limit of normal
* Creatinine =< 1.5 mg/dl OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Patients must have LVEF > 45%
* Patients must have baseline screening for G6PD (glucose-6-phosphate dehydrogenase) deficiency; G6PD must be no lower than the lower limit of normal prior to starting study treatment; patients who are above the upper limit of normal may enroll in the trial
* Patients must have measurable or evaluable disease
* The effects of Triapine® on the developing human fetus are unknown; for this reason and because heterocyclic carboxaldehyde thiosemicarbazones as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Patients who have not recovered from adverse events due to agents administered more than 4 weeks earlier; patients with grade =< 1 adverse events from prior therapies are eligible at the investigator's discretion
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Triapine® or other agents used in study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because Triapine® is a heterocyclic carboxaldehyde thiosemicarbazone with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Triapine®, breastfeeding should be discontinued if the mother is treated with Triapine®; these potential risks may also apply to other agents used in this study
* Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy; therefore, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with Triapine® or other agents administered during the study; appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated
* Patients with known G6PD deficiency are excluded
* Patients with severe pulmonary disease requiring oxygen and patients with baseline hypoxia (< 95% oxygen saturations) are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2004-01; Primary Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Number and severity of toxicity incidents categorized via Common Toxicity Criteria (CTC) standard toxicity grading | Up to 4 years
  Hematologic toxicity measures of thrombocytopenia, neutropenia and leukopenia will be assessed using the continuous variables as the outcome measures (primarily nadir and percent change from baseline values). Nonhematologic toxicities such as diarrhea and stomatitis will be evaluated via the ordinal CTC standard toxicity grading only. Frequency distributions and other descriptive measures will form the basis of the analysis of these variables.

SECONDARY OUTCOMES:
Number of responses | Up to 4 years
  Responses will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease.

CONTACTS AND LOCATIONS:
Overall Officials: George Wilding, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States